CLINICAL TRIAL: NCT02709291
Title: Systematically Adapted Delivery of the Family Check-Up in Underserved Communities
Brief Title: Systematically Adapted Delivery of the Family Check-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christina Studts (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Christina Studts, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R34MH106661 (NIH); R34MH106661 (NIH)
Record Dates: First submitted 2016-03-08; First posted 2016-03-16 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Parenting, Child Behavior, Implementation
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Workers (Other): Community health workers will complete a 5-day interventionist training to deliver a behavioral parent training intervention.
  Interventions: Behavioral: interventionist training
- Parent-Child Dyads (Other): Parents and children will receive a behavioral parent training intervention delivered by community health workers.
  Interventions: Behavioral: behavioral parent training

INTERVENTIONS:
Behavioral: behavioral parent training — Parents receive up to 6 sessions of the Family Check-Up program
  Arms: Parent-Child Dyads
Behavioral: interventionist training — Interventionists are trained in the delivery of the Family Check-Up program and deliver sessions to families in their community
  Arms: Community Health Workers

SUMMARY:
Early childhood disruptive behavior problems lead to significant costs to families and society, but can be reduced with behavioral parent training interventions. To increase the public health impact of these interventions, their feasibility, accessibility, and acceptability in high-need, underserved communities must be ensured. This pilot project will systematically adapt and pilot-test the delivery model of an existing effective parent training intervention for implementation in rural Appalachia, a region with many documented health disparities, high levels of poverty, and shortages of mental health providers. Community health workers in 5 rural Appalachian counties will be trained to deliver a behavioral parent training intervention. Each worker will deliver the intervention to 4 parent-child dyads.

ELIGIBILITY:
Inclusion Criteria:

* Parents: aged 18+ years, custodial guardian of child, can speak/read/understand English
* Children: ages 3-5 years, lives full time in custodial guardian's home
* Community health workers: aged 18+ years, currently employed at a partnering health department, able to speak/read/understand English

Exclusion Criteria:

* Parents: has already accessed behavioral health services for the child, reports suicidal ideation or intent to harm self or others, participated in formative research for this study
* Children: diagnosed with a severe developmental condition (i.e., significant developmental delay, autism, debilitating neurological condition)
* Community health workers: none

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Feasibility: Enrollment | 2 weeks after final parent-child dyad completes the study
  Percentage of invited parents who enroll in the study (obtained from process records)

SECONDARY OUTCOMES:
Feasibility: Number of sessions completed | 2 weeks after final parent-child dyad completes the study
  Number of sessions completed by each parent-child dyad (obtained from process records)
Feasibility: Interventionist-reported fidelity | following each behavioral parent training intervention session
  Fidelity Checklist (completed by community health workers)
Feasibility: Parent satisfaction | 10 weeks after parent baseline
  European Parent Satisfaction Scale about Early Intervention (EPASSEI) (completed by parents)
Interventionist satisfaction | 2 weeks after final parent-child dyad completes study
  Therapist Satisfaction Index (completed by community health workers)
Interventionist evidence-based practice attitudes | 2 weeks after final parent-child dyad completes study
  Evidence-Based Practice Attitude Scale-50 (completed by community health workers)
Interventionist self-efficacy | 2 weeks after final parent-child dyad completes study
  Counselor Activity Self-Efficacy Scale (completed by community health workers)

OTHER OUTCOMES:
Feasibility: Observer-rated fidelity | Throughout 10 weeks of behavioral parent training intervention per parent-child dyad
  Family Check-Up COACH fidelity rating system (observer-rated videos of 10% of intervention sessions)
Costs: Training | 2 weeks after final parent-child dyad completes study
  Total costs of training (obtained from process records maintained by investigators)
Costs: Per-family interventionist time | 2 weeks after final parent-child dyad completes study
  Obtained from process records maintained by community health workers
Costs: Per-family interventionist travel | 2 weeks after final parent-child dyad completes study
  Obtained from process records maintained by community health workers
Costs: Supervision time | 2 weeks after final parent-child dyad completes study
  Obtained from process records maintained by community health workers
Costs: Number of contacts outside of intervention sessions | 2 weeks after final parent-child dyad completes study
  Obtained from process records maintained by community health workers

CONTACTS AND LOCATIONS:
Overall Officials: Christina R Studts, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentuckyi, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No